CLINICAL TRIAL: NCT02001012
Title: Artemether-lumefantrine vs Chloroquine in Patients With Acute Uncomplicated P. Knowlesi Malaria: a Randomized Open Label Trial in Sabah, Malaysia (CAN KNOW Trial)
Brief Title: P. Knowlesi Trial of Artemether-lumefantrine vs Chloroquine
Acronym: CAN KNOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-13-18375
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Uncomplicated Knowlesi Malaria
Keywords: uncomplicated; plasmodium; knowlesi; malaria; infection
MeSH Terms: conditions — Malaria; Infections | interventions — Artemether, Lumefantrine Drug Combination; Chloroquine; Alkalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artemether-lumefantrine (Active Comparator): Artemether-lumefantrine.
  1 tablet = 20mg arthemether and 120mg lumefantrine. Dosing at 0, 8, 24, 36, 48 and 60 hours. Dose according to bodyweight; >35kg = 2 tablets, 26-35kg = 3 tablets, 16-25kg = 2 tablets, >10-15kg = 1 tablet.
  Interventions: Drug: Artemether-lumefantrine combination
- Chloroquine (Active Comparator): Chloroquine.
  1 tablet contains 155mg chloroquine base. Adult dose (>35kg); 620mg (4 tablets) at 0 hours, and 310mg (2 tablets) at 6-8, 24 and 48 hours.
  Child dose (>10-35kg); 10mg/kg at 0 hours, and 5mg/kg at 6-8, 24 and 48 hours.
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Artemether-lumefantrine combination
  Other Names: Riamet; Co-Artem
  Arms: Artemether-lumefantrine
Drug: Chloroquine
  Other Names: Chloroquine; 1 tablet = 155mg base
  Arms: Chloroquine

SUMMARY:
Preliminary studies have supported the background efficacy of local standard anti-malarial medications in the treatment of uncomplicated knowlesi malaria, however there are no current WHO treatment guidelines for this infection. There are both health cost benefits to a more rapidly acting agent, and due to difficulties with microscopic identification there may be more effective treatment for all malaria species if an aligned treatment guideline could be supported. We are currently conducting a separate RCT using a similar protocol evaluating artesunate-mefloquine versus chloroquine for uncomplicated P. knowlesi malaria. However artemether-lumefantrine should also be compared against chloroquine due to the fact it is also a first line anti-malarial recommended in Malaysia, and there are potential differences in efficacy due to the different administration, absorption and half-life of artemether-lumefantrine.

The investigators aim to test whether the fixed combination of artesunate-mefloquine is superior to chloroquine in order to define the optimal treatment for both uncomplicated P. knowlesi infection in both adults and children in this region.

DETAILED DESCRIPTION:
Naturally acquired infections with Plasmodium knowlesi, the fifth human malaria, are growing [1]. Since 2004 increasing numbers of cases have been reported from residents and returned travelers predominantly from Malaysia and other countries in South-East Asia including Thailand, Vietnam, Myanmar, Singapore, Indonesia and the Philippines [2-8]. Cases coincide with the geographic distribution of its natural simian hosts (long-tailed and pig-tailed macaques) and Anopheles leucosphyrus group mosquito vector [9, 10], with potential human-to-human transmission unknown. Eastern Malaysia appears to be the epicentre, with around 1400 PCR-confirmed P. knowlesi human mono-infections reported in 2009, comprising 41% of 2,189 total malaria cases in Sarawak [11] and 343 cases from selected samples sent to Sabah's State Reference Laboratory [12]. P. knowlesi is also now the most common cause of malaria in different contrasting regions, including 70% of malaria admissions in the heavily forested area of Kapit in Sarawak [1, 13], 63% of samples from the interior division of Sabah [14], and in 87% of malaria admissions in the deforested coastal area of Kudat in Sabah, where it is also the major cause of malaria in children [15].

Despite the increase in reported incidence, difficulties with microscopic diagnosis and a lack of PCR based epidemiological surveillance studies throughout South-East Asia mean the true disease burden is underestimated. P. knowlesi is microscopically misidentified as P . falciparum and P. malariae due to morphological similarities in the early trophozoite, and late trophozoite and schizont life stages respectively, with studies showing up to 80% of P. malariae [16-19] and 7-12% of P. falciparum [1, 16] in this region are actually P. knowlesi when definitively evaluated with PCR. Misdiagnosis has concerning treatment implications, as unlike P. malariae, knowlesi malaria has a rapid 24-hour replication rate and can cause hyperparasitaemia, severe complications and fatal outcomes [13, 17, 18], while the inadvertent use of chloroquine for widely chloroquine-resistant P. falciparum may also have fatal consequences.

Naturally acquired infections with Plasmodium knowlesi, the fifth human malaria, are growing [1]. Since 2004 increasing numbers of cases have been reported from residents and returned travelers predominantly from Malaysia and other countries in South-East Asia including Thailand, Vietnam, Myanmar, Singapore, Indonesia and the Philippines [2-8]. Cases coincide with the geographic distribution of its natural simian hosts (long-tailed and pig-tailed macaques) and Anopheles leucosphyrus group mosquito vector [9, 10], with potential human-to-human transmission unknown. Eastern Malaysia appears to be the epicentre, with around 1400 PCR-confirmed P. knowlesi human mono-infections reported in 2009, comprising 41% of 2,189 total malaria cases in Sarawak [11] and 343 cases from selected samples sent to Sabah's State Reference Laboratory [12]. P. knowlesi is also now the most common cause of malaria in different contrasting regions, including 70% of malaria admissions in the heavily forested area of Kapit in Sarawak [1, 13], 63% of samples from the interior division of Sabah [14], and in 87% of malaria admissions in the deforested coastal area of Kudat in Sabah, where it is also the major cause of malaria in children [15].

Despite the increase in reported incidence, difficulties with microscopic diagnosis and a lack of PCR based epidemiological surveillance studies throughout South-East Asia mean the true disease burden is underestimated. P. knowlesi is microscopically misidentified as P . falciparum and P. malariae due to morphological similarities in the early trophozoite, and late trophozoite and schizont life stages respectively, with studies showing up to 80% of P. malariae [16-19] and 7-12% of P. falciparum [1, 16] in this region are actually P. knowlesi when definitively evaluated with PCR. Current rapid diagnostic tests (RDT) for malaria can distinguish falciparum Current rapid diagnostic tests (RDT) for malaria can distinguish falciparum from other Plasmodium species with a sensitivity of up to 99% at parasite counts > 1,000/ μL [20], but a knowlesi specific antigen has not been developed and current antibody panels are unable to differentiate between P. knowlesi and other mixed Plasmodium spp. infections [21]. Misdiagnosis has concerning treatment implications, as unlike P. malariae, knowlesi malaria has a rapid 24-hour replication rate and can cause hyperparasitaemia, severe complications and fatal outcomes [13, 17, 18], while the inadvertent use of chloroquine for widely chloroquine-resistant P. falciparum may also have fatal consequences.

Artemether-lumefantrine (A-L) is a common and widely available ACT, and along with artesunate-mefloquine (AS-MQ) is one of only 2 first line WHO recommended options for the treatment of uncomplicated P.falciparum infection which are registered in Malaysia and produced according to international good manufacturing practice (GMP) standards. ACTs are the current mainstay of malaria eradication efforts 28, with a mechanism of action resulting both in a rapid reduction in parasite mass and resolution of clinical features, while the long acting component eliminates residual parasites and delays the development of de novo resistance 29,30.

Initial reported use of A-L for knowlesi malaria was from our retrospective study at a tertiary referral hospital in Sabah, where a small sample size of 8 out of 34 patients with PCR confirmed uncomplicated P.knowlesi infection were treated with oral artemether-lumefantrine. Median microscopic parasite clearance time was 1 day (range 0-3), which was significantly faster than those receiving chloroquine (median 2.5 days, range 1-3), while this also resulted in fewer days of hospitalization and health sector associated costs. The proportion remaining parasitaemic at day 1 was 33% 16. Our subsequent prospective study at the same site documented 109 knowlesi malaria patients successfully treated with A-L, with no recurrences identified. Unpublished data from this study showed that of the patients with uncomplicated P. knowlesi malaria enrolled, 51 received A-L monotherapy, with a median parasite clearance time of 2 days31.

Evaluation of A-L is required in addition to AS-MQ, as there are a number of pharmacokinetic and pharmacodynamic differences that may affect clinical outcomes. In contrast to AS-MQ, adequate oral absorption of A-L requires co-adminstration with fatty foods, with twice daily dosing28. The longer acting partner drug in A-L is lumefantrine, which has a half life of 3 days compared to mefloquine in AS-MQ which is 21 days. Therefore there may be differences in P. knowlesi recurrence at day 28 or 42 as the follow up time recommended by WHO for anti-malarial efficacy monitoring studies 32.

Chloroquine with primaquine was initially suggested to have favourable treatment outcomes for uncomplicated P. knowlesi human infections after a retrospective review of patients from Kapit Hospital in Sarawak in 2004 15. Following this a single prospective observational study conducted at the same site between 2006-7 administered chloroquine as a total base dose of 25mg/kg and primaquine as a gametocidal agent to 73 patients with uncomplicated PCR-confirmed P. knowlesi malaria, with results showing median fever clearance of 26 hours, mean times to 50% and 90% microscopic parasite clearance of 3.1 and 10.3 hours respectively, and a median PCR adjusted clearance time of 3 days. The proportion remaining parasitaemic at day 1 was 55%. None of the 60 patients who completed the 28-day follow up demonstrated any evidence of resistance, re-infection or recrudescence 25.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 1 year of age and weighing more than 10kg.
* Microscopic diagnosis P. knowlesi (including diagnosis as P. malariae) or P. falciparum infection (any parasitaemia).
* Negative P. falciparum malaria rapid diagnostic test (histidine rich protein 2)
* Fever (temperature ≥37.5°C) or history of fever in the last 48 hours.
* Able to participate in the trial and comply with the clinical trial protocol.
* Written informed consent to participate in trial; thumbprint is required for illiterate patients, and written consent from parents/guardian for children below age of consent.

Exclusion Criteria:

* Clinical or laboratory criteria for severe malaria, including warning signs, requiring parenteral treatment according to modified WHO criteria (see Appendix 4)
* Parasitaemia > 20,000 /μL
* Inability to tolerate oral treatment
* Concomitant infection with any other malaria species
* Positive for P. falciparum histidine-rich-protein-2 by malaria rapid diagnostic test
* Pregnancy or lactation
* Unable or unwilling to use contraception during study period
* Known hypersensitivity or allergy to artemisinin derivatives
* Serious underlying disease (cardiac, renal or hepatic)
* Received anti-malarials in previous 2 months
* Previous psychiatric illness or epilepsy
* Previous episode of cerebral malaria

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Parasite clearance | 24 hours
  The primary endpoint is the therapeutic efficacy of artemether-lumefantrine versus chloroquine, as defined by the assessment of microscopic P. knowlesi parasite clearance 24 hours after initiation of treatment.

SECONDARY OUTCOMES:
Rates of recurrent infection / treatment failure at day 42. | 42 days
Occurrence of anaemia at day 28 when using AL vs. CQ. | 28 days
P. knowlesi and gametocyte carriage throughout follow up when using AL vs. CQ. | 42 days
Frequency of complications throughout follow up when using AL vs. CQ. | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Jayaram Menon, MBBS, Study Director — Sabah Ministry of Health; Matthew Grigg, MBBS, Study Director — Menzies School of Health Research; Prabakaran Dhanaraj, MBBS, Study Director — Sabah Ministry of Health; Tsin Yeo, MBBS, Study Director — Menzies School of Health Research; Bridget Barber, MBBS, Study Director — Menzies School of Health Research; Nicholas Anstey, MBBS, Study Director — Menzies School of Health Research; Ric Price, MBBS, Study Director — Menzies School of Health Research
Locations (3):
- Malaysia (3):
  - Kota Marudu District Hospital, Kota Marudu, Sabah
  - Kudat District Hospital, Kudat, Sabah
  - Pitas District Hospital, Pitas, Sabah

REFERENCES:
- [Background] Cox-Singh J, Davis TM, Lee KS, Shamsul SS, Matusop A, Ratnam S, Rahman HA, Conway DJ, Singh B. Plasmodium knowlesi malaria in humans is widely distributed and potentially life threatening. Clin Infect Dis. 2008 Jan 15;46(2):165-71. doi: 10.1086/524888. PMID 18171245
- [Background] Putaporntip C, Hongsrimuang T, Seethamchai S, Kobasa T, Limkittikul K, Cui L, Jongwutiwes S. Differential prevalence of Plasmodium infections and cryptic Plasmodium knowlesi malaria in humans in Thailand. J Infect Dis. 2009 Apr 15;199(8):1143-50. doi: 10.1086/597414. PMID 19284284
- [Background] Marchand RP, Culleton R, Maeno Y, Quang NT, Nakazawa S. Co-infections of Plasmodium knowlesi, P. falciparum, and P. vivax among Humans and Anopheles dirus Mosquitoes, Southern Vietnam. Emerg Infect Dis. 2011 Jul;17(7):1232-9. doi: 10.3201/eid1707.101551. PMID 21762577
- [Background] Ng OT, Ooi EE, Lee CC, Lee PJ, Ng LC, Pei SW, Tu TM, Loh JP, Leo YS. Naturally acquired human Plasmodium knowlesi infection, Singapore. Emerg Infect Dis. 2008 May;14(5):814-6. doi: 10.3201/eid1405.070863. PMID 18439370
- [Background] Luchavez J, Espino F, Curameng P, Espina R, Bell D, Chiodini P, Nolder D, Sutherland C, Lee KS, Singh B. Human Infections with Plasmodium knowlesi, the Philippines. Emerg Infect Dis. 2008 May;14(5):811-3. doi: 10.3201/eid1405.071407. PMID 18439369
- [Background] Singh B, Daneshvar C. Plasmodium knowlesi malaria in Malaysia. Med J Malaysia. 2010 Sep;65(3):166-72. PMID 21939162
- [Derived] Grigg MJ, William T, Barber BE, Rajahram GS, Menon J, Schimann E, Wilkes CS, Patel K, Chandna A, Price RN, Yeo TW, Anstey NM. Artemether-Lumefantrine Versus Chloroquine for the Treatment of Uncomplicated Plasmodium knowlesi Malaria: An Open-Label Randomized Controlled Trial CAN KNOW. Clin Infect Dis. 2018 Jan 6;66(2):229-236. doi: 10.1093/cid/cix779. PMID 29020373